CLINICAL TRIAL: NCT00938158
Title: An Adaptive Design Study for the Assessment of the Pharmacokinetics of Albiglutide in Subjects With Normal Renal Function and Subjects With Moderate-to-severe Renal Impairment and Hemodialysis.
Brief Title: A Study of the Pharmacokinetics of Albiglutide in Normal and Renally Impaired Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108370
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: albiglutide; hemodialysis; pharmacokinetics; renal
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Stage 1 normal renal function (Experimental): Subject with estimated glomerular filtration rate (GFR) greater than 80 milliliter per minute (mL/min)
  Interventions: Biological: albiglutide
- Stage 1 moderate/severe renal function (Experimental): Subject with estimated GFR >= 20 mL/min and less than 50 mL/min
  Interventions: Biological: albiglutide
- Stage 2 normal renal function (Experimental): Subject with GFR greater than 80 mL/min
  Interventions: Biological: albiglutide
- Stage 2 moderate renal impairment (Experimental): Subject with estimated GFR >= 30 mL/min and less than 50 mL/min
  Interventions: Biological: albiglutide
- Stage 2 subjects requiring hemodialysis (Experimental): Subjects who require hemodialysis
  Interventions: Biological: albiglutide
- Stage 2 severe renal impairment not requiring hemodialysis (Experimental): Subjects with GFR less than 30 mL/min
  Interventions: Biological: albiglutide
- Stage 2 mild renal impairment (Experimental): Subjects with GFR >= 50 mL/min and <= 80 mL/min
  Interventions: Biological: albiglutide

INTERVENTIONS:
Biological: albiglutide — single dose of subcutaneously injected albiglutide

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of a single subcutaneously injected dose of albiglutide in subjects with type 2 diabetes mellitus with varying degrees of renal function, including subjects requiring hemodialysis.

DETAILED DESCRIPTION:
This adaptive design, non-randomized, open-label, staggered parallel group study evaluates the pharmacokinetics and safety of a single subcutaneously injected dose of albiglutide in subjects with type 2 diabetes mellitus with varying degrees of renal function. During Stage 1, a single dose of albiglutide will be administered to subjects with normal renal function and subjects with moderate-to-severe renal impairment not requiring hemodialysis. In addition to subjects with normal renal function and moderate renal impairment, Stage 2 of the study will also include cohorts of subjects requiring hemodialysis, subjects with severe renal impairment not requiring hemodialysis, and potentially subjects with mild renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* normal renal function or renal impairment
* stable hemodialysis treatment for at least 3 months before screening and able to tolerate a hemodialysis treatment lasting 3-4 hours with blood flow rates of >200mL/min (cohort 3 only)
* neither pregnant nor lactating
* HbA1c 6-10.5% inclusive
* females of childbearing potential must be practicing adequate contraception.

Exclusion Criteria:

* inability to meet the PK objectives of the study
* history of hypoglycemia unawareness or severe hypoglycemia
* liver function tests greater than or equal to 2 times the ULN
* clinically significant cardiovascular and/or cerebrovascular disease
* positive test results for hepatitis B, hepatitis C, or HIV
* documented hypertension or hypotension at screening
* known hepatic or biliary abnormalities
* current use of sulfonylureas
* active history of tobacco use within 6 months before screening
* donation of blood in excess of 500mL within 56 days before albiglutide dosing
* receipt of any investigational drug within the 30days or 5 half lives, whichever is longer, before dosing
* previous or current receipt of exenatide or any other GLP-1 agonist

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-08-05 (Actual); Primary Completion 2011-04-12 (Actual); Study Completion 2011-04-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to characterize the PK of albiglutide in subjects with type 2 diabetes and varying degrees of renal impairment, including subjects requiring hemodialysis, and in age, gender and BMI-matched subjects. | 42 days

SECONDARY OUTCOMES:
To assess the PK of albiglutide in subjects with varying degrees of proteinuria | 42 days
To assess the effects of hemodialysis on the overall PK profile of albiglutide | 42 days
To assess the safety and tolerability of a single dose of albiglutide in subjects with varying degrees of renal impairment and in age, gender and BMI-matched subjects with normal renal function | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (5):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Minneapolis, Minnesota
- South Africa (2):
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Somerset West

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- [Derived] Young MA, Wald JA, Matthews JE, Yang F, Reinhardt RR. Effect of renal impairment on the pharmacokinetics, efficacy, and safety of albiglutide. Postgrad Med. 2014 May;126(3):35-46. doi: 10.3810/pgm.2014.05.2754. PMID 24918790
- See also: Results for study 108370 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/108370?search=study&search_terms=108370#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 108370 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108370 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108370 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108370 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108370 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108370 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108370 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register